CLINICAL TRIAL: NCT02413281
Title: A Phase 1, Single-Dose, Double-Blind, Placebo-and Active-Controlled, Randomized, 6-way Crossover Human Abuse Liability Evaluation of ALKS 5461
Brief Title: A Study of the Abuse Liability Potential of ALKS 5461 in Healthy, Non-Dependent, Recreational Opioid Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ALK5461-212
Record Dates: First submitted 2015-04-07; First posted 2015-04-09 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Healthy Volunteer; Abuse Liability; ALKS 5461; Alkermes
MeSH Terms: interventions — ALKS 5461; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- ALKS 5461 Dose 1 (Experimental): Sublingual tablets
  Interventions: Drug: ALKS 5461
- ALKS 5461 Dose 2 (Experimental): Sublingual tablets
  Interventions: Drug: ALKS 5461
- ALKS 5461 Dose 3 (Experimental): Sublingual tablets
  Interventions: Drug: ALKS 5461
- Buprenorphine Dose 1 (Active Comparator): Sublingual tablets
  Interventions: Drug: Buprenorphine
- Buprenorphine Dose 2 (Active Comparator): Sublingual tablets
  Interventions: Drug: Buprenorphine
- Placebo (Placebo Comparator): Sublingual tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 5461 — Sublingual tablets, single administration
  Arms: ALKS 5461 Dose 1; ALKS 5461 Dose 2; ALKS 5461 Dose 3
Drug: Buprenorphine — Sublingual tablets, single administration
  Arms: Buprenorphine Dose 1; Buprenorphine Dose 2
Drug: Placebo — Sublingual tablets, single administration
  Arms: Placebo

SUMMARY:
This study will evaluate the abuse potential of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) within the range of 18.0 to 30.0 kg/m2, inclusive, and a minimum weight of at least 50.0 kg
* Be a current recreational opioid user who has used opioids for non-therapeutic purposes (ie for psychoactive effects) at least 10 times in their lifetime
* Agree to use an approved method of contraception for the duration of the study unless surgically sterile or postmenopausal
* Be willing and able to abide by all study requirements and restrictions
* Additional criteria may apply

Exclusion Criteria:

* Have evidence of drug or alcohol dependence within the past 2 years
* Have a positive drug screen for opioids, amphetamines, cocaine, or benzodiazepines upon admission to the clinic
* Have a history of severe allergic reaction (including anaphylaxis) to any food, medication, or bee sting
* Be currently pregnant, breastfeeding, or planning to become pregnant during the study
* Currently have or have a history of allergy or hypersensitivity to opioid agonists, opioid antagonists or related drugs (eg, oxycodone, morphine, naltrexone, and naloxone)
* Have a positive test result for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Have donated or lost more than 500 mL whole blood
* Additional criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: Abuse potential measured by visual analog scales (VAS) | Approximately 14 weeks

SECONDARY OUTCOMES:
Safety: Incidence of adverse events (AEs) | Up to 14 weeks
Pharmacokinetics: Plasma concentrations of ALKS 5461 | Up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Pathak S, Vince B, Kelsh D, Shram MJ, Setnik B, Lu H, Nangia N, Stanford AD, Ehrich E. Abuse Potential of Buprenorphine/Samidorphan Combination Compared to Buprenorphine and Placebo: A Phase 1 Randomized Controlled Trial. J Clin Pharmacol. 2019 Feb;59(2):206-217. doi: 10.1002/jcph.1280. Epub 2018 Aug 13. PMID 30102427